CLINICAL TRIAL: NCT05966805
Title: Examining the Impact of a 12-week Worksite Exercise Training Intervention on Mental, Metabolic, Physical, Spiritual, and Occupational Well-being Among Acute Care Nurses: A Randomized, Controlled Mixed Methods Pilot Study
Brief Title: Impact of Exercise Intervention on Well-being in Shift-working Acute Care Nurses
Acronym: WELL_NURSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1762353
Record Dates: First submitted 2023-06-06; First posted 2023-08-01 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-09

CONDITIONS: Psychological Wellness
Keywords: exercise; whole person health; nurses; pilot study
MeSH Terms: conditions — Psychological Well-Being; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training Group (Experimental): Exercise intervention group will undergo a 12-week exercise program.
  Interventions: Behavioral: Exercise training group
- Wait-List Control Group (Other): Wait-List control group will participate in visits every 4 weeks for data collection and periodic phone calls for monitoring. They will be offered the exercise training intervention option at conclusion.
  Interventions: Behavioral: Wait-List Control Group

INTERVENTIONS:
Behavioral: Exercise training group — 12-Week Exercise intervention on mentaL, metabolic, physicaL, spiritual, social, and occupational well-being among shift-working acute care NURSE
  Arms: Exercise Training Group
Behavioral: Wait-List Control Group — Control group
  Arms: Wait-List Control Group

SUMMARY:
This is a randomized, wait-list control pilot study to analyze the impact of a 12-week exercise training intervention on post-traumatic growth and whole-person well-being (mental health, physical health, spiritual well-being, perceived social support, and occupational health) among shift-working acute care nurses within AdventHealth.

DETAILED DESCRIPTION:
This study has five phases: Phase I: Screening; Phase II: Baseline Assessments (Pre-Intervention); Phase III: Exercise training; Phase IV: Post-Intervention; and Phase V: Repeat assessments at 3-months and 6-months post-intervention.

Phase I (90 minutes): This phase consists of reviewing and obtaining consent, screening for inclusion/exclusion criteria, reviewing study details, and assessing the need for medical clearance to participate in the exercise intervention, and a single blood draw for fasted blood profiles.

Phase II (7 hours): Upon successful screening, all participants will complete baseline assessments.

Phase III (Exercise Training Group 34 hours/Wait-List Control 4.5 hours): Upon completion of Phase II, participants will be randomized to the exercise training intervention group or the wait-list control group.

Phase IV (7 hours): All participants will enter a post-intervention phase that includes repeat assessments of Phase II outcomes.

Phase V (~2 hours): A subset of psychometric questionnaires will be repeated 3- and 6-months post-exercise training intervention to ascertain sustainability of the intervention.

*Subjects randomized to the wait-list control group will be offered the exercise training intervention upon completion of the Phase V assessments.

ELIGIBILITY:
Inclusion:

1. Age 21-65 years
2. Nurse working in an AdventHealth inpatient acute care setting
3. Currently working as a shift-working acute care nurse within AdventHealth.
4. Weight stable prior to beginning the study exercise training intervention.
5. Able to speak and understand written and spoken English.
6. Understands the procedures and agrees to participate by giving written informed consent.
7. Willing and able to comply with scheduled visits, laboratory tests, and other study procedures including a 12-week exercise training program.

Exclusion Criteria:

1. Positive urine pregnancy test prior to DEXA scan
2. Uncontrolled Type 1 or Type 2 diabetes mellitus
3. Bleeding disorders
4. Acute or chronic infections
5. Chronic obstructive pulmonary disease
6. Renal insufficiency or nephritis
7. Uncontrolled hypertension (BP>160 mmHg systolic or >100 mmHg diastolic)
8. History of Cushing's disease or syndrome
9. Active rheumatoid arthritis or other inflammatory rheumatic disorder
10. Major surgery within 4 weeks prior to Screening
11. Participation in studies involving investigational drug(s) within 30 days prior to Screening
12. History or presence of cardiovascular disease (unstable angina, myocardial infarction or coronary revascularization within 6 months, presence of cardiac pacemaker, implanted cardiac defibrillator)
13. Any malignancy not considered cured, except basal cell carcinoma and squamous cell carcinoma of the skin (a participant is considered cured if there has been no evidence of cancer recurrence in the previous 5 years)
14. Presence of any condition that, in the opinion of the Investigator or medical investigator, compromises participant safety or data integrity or the participant's ability to complete study days.
15. More than 1-day a week of intentional exercise
16. Medically diagnosed sleep disorder
17. Weight >450 lbs

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Post-traumatic growth | Group comparison baseline, 3 months, and 6 months follow-up
  Post-traumatic growth inventory (PTGI) (21-item questionnaire with Likert scale of 0-5, with 0 for "I did not experience this change as a result of my crisis" and 5 for "I experienced this change to a very great degree as a result of my crisis")

SECONDARY OUTCOMES:
Depression | Group comparisons baseline, 3 months, and 6 months follow-up
  Patient Health Questionnaire (PHQ-2) (2-items measuring depression using Likert scale of 0 to 3 with 0 for "not at all" and 3 for "nearly every day)
Anxiety | Group comparisons baseline, 3 months, and 6 months follow-up
  Generalized Anxiety Disorder Scale (GAD-2) (2-items measuring anxiety with 4-point Likert scale with 0 for "not at all" and 3 for "nearly every day")
Professional Quality of Life for Health care workers | Group comparisons baseline, 3 months, and 6 months follow-up
  Professional Quality of Life Health (Pro-QOL Health) (30-items covering five domains (6 items each domain): 1) Compassion Satisfaction, 2) Perceived Support, 3) Burnout, 4) Secondary Traumatic Stress, and 5) Moral Distress using a Likert scale of 1-5 with 1 for "never" and 5 for "very often")
Cardiorespiratory fitness | Group comparisons baseline, 3 months follow-up
  Cardiopulmonary exercise test (CPX-T). (Aerobic fitness will be determined by measuring maximal O2 consumption (VO2max) during a stationary bicycle test)
24-H Physical activity patterns | Group comparisons baseline, 3 months follow-up
  GT3-X-BT, ActiGraph, LLC) monitor integrates motion sensor data from the tri-axial accelerometer to estimate the energy cost of free-living activity
Spiritual well-being | Group comparisons baseline, 3 months, and 6 months follow-up
  FACIT Spiritual Well-Being (FACIT-Sp) Non-Illness Version (12-items with a 5-point Likert with total score range from 0-32 with higher scores indicating better QOL/spiritual well-being)
Job Satisfaction | Group comparisons baseline, 3 months, and 6 months follow-up
  Nurse Job Satisfaction Scale (7 items using a 5-point Likert scale from 1 for "strongly disagree" to 5 for "strongly agree")
Missed Care | Group comparisons baseline, 3 months, and 6 months follow-up
  NDNQI Index of Work Satisfaction missed care (Two multiple choice questions about the last shift worked)
Work-related exhaustion | Group comparisons baseline, 3 months, and 6 months follow-up
  Quality Work Competence (3-item subscale with 5-point Likert scale from 1 for "never" to 5 for "very often")
Medical Errors | Group comparisons baseline, 3 months, and 6 months follow-up
  Single-item medical error question.
Sleep | Group comparisons baseline, week 12
  GT3-X-BT, ActiGraph, LLC) monitor integrates motion sensor data from the tri-axial accelerometer sleep measurements to determine total sleep time, sleep efficiency, and sleep latency.
Sleep questionnaire | Group comparisons baseline, week 12
  Morningness-eveningness questionnaire Self-Report version (MEQ-REV-SR) (4 multiple choice items)
Sleep diary | Group comparisons baseline, week 12
  National sleep foundation 7-day sleep diary (7 items for am and 8 items for pm)
Cognitive Health | Group comparison baseline, 1 week follow-up
  Workplace Cognitive Failure Scale (15 items about experiences during last work week with Likert scale from 1 for "never" to 5 for "very often")
Insulin resistance | Group comparison baseline, 1 week follow-up
  Blood collection fasting glucose, fasting insulin, lipid panel profile
Weight | Group comparison baseline, week 1, week 4, week 8, week 12, 1 week follow-up
  Weight in kilograms
Waist circumference | Group comparison baseline, week 1, week 4, week 8, week 12, 1 week follow-up
  Waist circumference in centimeters
Body Mass Index | Group comparison baseline, week 1, week 4, week 8, week 12, 1 week follow-up
  Calculated body mass index based on current weight in kilograms and height in centimeters taken at baseline
Body composition | Group comparison baseline, 1 week follow-up
  DEXA scan
Nutrition | Group comparison baseline, 1 week follow-up
  Diet history Questionnaire-III (DHQ-III) (A questionnaire on beverage and food intake over the past month with branching items on amount of consumption based on responses)
Physical condition - strength | Group comparison baseline, 1 week follow-up
  Muscle power testing will be performed using a Biodex pneumatic-driven dynamometer
Physical Activity | Group comparison baseline, 1 week follow-up
  International Physical Activity Questionnaire (IPAQ) (27 maximum branching items with 5 parts: 1) Job-related physical activity, 2) Transportation physical activity, 3) Housework, house maintenance, and caring for family, 4) Recreation, sport, and leisure-time physical activity, 5) Time spent sitting
Lifestyle Beliefs | Group comparison baseline, 1 week follow-up
  Healthy Lifestyle Beliefs Scale (16 items with 5-point Likert scale from "Strongly Disagree" to "Strongly Agree"
Lifestyle Behaviors | Group comparison baseline, 1 week follow-up
  Healthy Lifestyle Behaviors Scale (16 items with 5-point Likert scale from "Strongly Disagree" to "Strongly Agree"

OTHER OUTCOMES:
Adherence/Compliance | 1 week follow-up
  Percentage of exercise session attendance (number of attended sessions/the number of scheduled sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Brennan, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gan Y, Yang C, Tong X, Sun H, Cong Y, Yin X, Li L, Cao S, Dong X, Gong Y, Shi O, Deng J, Bi H, Lu Z. Shift work and diabetes mellitus: a meta-analysis of observational studies. Occup Environ Med. 2015 Jan;72(1):72-8. doi: 10.1136/oemed-2014-102150. Epub 2014 Jul 16. PMID 25030030
- [Background] Gu F, Han J, Laden F, Pan A, Caporaso NE, Stampfer MJ, Kawachi I, Rexrode KM, Willett WC, Hankinson SE, Speizer FE, Schernhammer ES. Total and cause-specific mortality of U.S. nurses working rotating night shifts. Am J Prev Med. 2015 Mar;48(3):241-52. doi: 10.1016/j.amepre.2014.10.018. Epub 2015 Jan 6. PMID 25576495
- [Background] Vetter C, Devore EE, Wegrzyn LR, Massa J, Speizer FE, Kawachi I, Rosner B, Stampfer MJ, Schernhammer ES. Association Between Rotating Night Shift Work and Risk of Coronary Heart Disease Among Women. JAMA. 2016 Apr 26;315(16):1726-34. doi: 10.1001/jama.2016.4454. PMID 27115377
- [Background] Brown JP, Martin D, Nagaria Z, Verceles AC, Jobe SL, Wickwire EM. Mental Health Consequences of Shift Work: An Updated Review. Curr Psychiatry Rep. 2020 Jan 18;22(2):7. doi: 10.1007/s11920-020-1131-z. PMID 31955278
- [Background] Torquati L, Mielke GI, Brown WJ, Burton NW, Kolbe-Alexander TL. Shift Work and Poor Mental Health: A Meta-Analysis of Longitudinal Studies. Am J Public Health. 2019 Nov;109(11):e13-e20. doi: 10.2105/AJPH.2019.305278. Epub 2019 Sep 19. PMID 31536404
- [Background] American Nurses Association. Healthy Nurse Healthy Nation: Year Three Highlights 2019-2020, <https://www.healthynursehealthynation.org/globalassets/all-images-view-with-media/about/2020-hnhn_sup-8.pdf> (2020)
- [Background] Chellappa SL, Morris CJ, Scheer FAJL. Circadian misalignment increases mood vulnerability in simulated shift work. Sci Rep. 2020 Oct 29;10(1):18614. doi: 10.1038/s41598-020-75245-9. PMID 33122670
- [Background] Scheer FAJL, Chellappa SL, Hu K, Shea SA. Impact of mental stress, the circadian system and their interaction on human cardiovascular function. Psychoneuroendocrinology. 2019 May;103:125-129. doi: 10.1016/j.psyneuen.2019.01.016. Epub 2019 Jan 16. PMID 30682628
- [Background] Sletten TL, Cappuccio FP, Davidson AJ, Van Cauter E, Rajaratnam SMW, Scheer FAJL. Health consequences of circadian disruption. Sleep. 2020 Jan 13;43(1):zsz194. doi: 10.1093/sleep/zsz194. No abstract available. PMID 31930347
- [Background] Vetter C, Scheer FAJL. A healthy lifestyle - reducing T2DM risk in shift workers? Nat Rev Endocrinol. 2019 Apr;15(4):194-196. doi: 10.1038/s41574-019-0164-z. No abstract available. PMID 30718862
- [Background] McHill AW, Melanson EL, Higgins J, Connick E, Moehlman TM, Stothard ER, Wright KP Jr. Impact of circadian misalignment on energy metabolism during simulated nightshift work. Proc Natl Acad Sci U S A. 2014 Dec 2;111(48):17302-7. doi: 10.1073/pnas.1412021111. Epub 2014 Nov 17. PMID 25404342
- [Background] Stuijfzand S, Deforges C, Sandoz V, Sajin CT, Jaques C, Elmers J, Horsch A. Psychological impact of an epidemic/pandemic on the mental health of healthcare professionals: a rapid review. BMC Public Health. 2020 Aug 12;20(1):1230. doi: 10.1186/s12889-020-09322-z. PMID 32787815
- [Background] Hall LH, Johnson J, Watt I, Tsipa A, O'Connor DB. Healthcare Staff Wellbeing, Burnout, and Patient Safety: A Systematic Review. PLoS One. 2016 Jul 8;11(7):e0159015. doi: 10.1371/journal.pone.0159015. eCollection 2016. PMID 27391946
- [Background] Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports. 2015 Dec;25 Suppl 3:1-72. doi: 10.1111/sms.12581. PMID 26606383
- [Background] Melnyk BM, Kelly SA, Stephens J, Dhakal K, McGovern C, Tucker S, Hoying J, McRae K, Ault S, Spurlock E, Bird SB. Interventions to Improve Mental Health, Well-Being, Physical Health, and Lifestyle Behaviors in Physicians and Nurses: A Systematic Review. Am J Health Promot. 2020 Nov;34(8):929-941. doi: 10.1177/0890117120920451. Epub 2020 Apr 27. PMID 32338522
- [Background] Bischoff LL, Otto AK, Hold C, Wollesen B. The effect of physical activity interventions on occupational stress for health personnel: A systematic review. Int J Nurs Stud. 2019 Sep;97:94-104. doi: 10.1016/j.ijnurstu.2019.06.002. Epub 2019 Jun 11. PMID 31234106
- [Background] Chappel SE, Verswijveren SJJM, Aisbett B, Considine J, Ridgers ND. Nurses' occupational physical activity levels: A systematic review. Int J Nurs Stud. 2017 Aug;73:52-62. doi: 10.1016/j.ijnurstu.2017.05.006. Epub 2017 May 10. PMID 28535398
- [Background] Chen, J. et al. Physical activity and post-traumatic growth: A systematic review of quantitative and qualitative studies. Psychology of Sport & Exercise 49, doi:10.1016/j.psychsport.2020.101679 (2020).
- [Background] Constandt B, Thibaut E, De Bosscher V, Scheerder J, Ricour M, Willem A. Exercising in Times of Lockdown: An Analysis of the Impact of COVID-19 on Levels and Patterns of Exercise among Adults in Belgium. Int J Environ Res Public Health. 2020 Jun 10;17(11):4144. doi: 10.3390/ijerph17114144. PMID 32532013
- [Background] Coulson, J. C., McKenna, J. & Field, M. Exercising at work and self-reported work performance. International Journal of Workplace Health Management 1, 176-197, doi:10/1108/17538350810926534 (2008).
- [Background] Doran K, Resnick B, Alghzawi H, Zhu S. The worksite heart health improvement project's impact on behavioral risk factors for cardiovascular disease in long-term care: A randomized control trial. Int J Nurs Stud. 2018 Oct;86:107-114. doi: 10.1016/j.ijnurstu.2018.06.011. Epub 2018 Jun 28. PMID 30005312
- [Background] Jakobsen MD, Sundstrup E, Brandt M, Andersen LL. Psychosocial benefits of workplace physical exercise: cluster randomized controlled trial. BMC Public Health. 2017 Oct 10;17(1):798. doi: 10.1186/s12889-017-4728-3. PMID 29017479
- [Background] Matsugaki R, Kuhara S, Saeki S, Jiang Y, Michishita R, Ohta M, Yamato H. Effectiveness of workplace exercise supervised by a physical therapist among nurses conducting shift work: A randomized controlled trial. J Occup Health. 2017 Jul 27;59(4):327-335. doi: 10.1539/joh.16-0125-OA. Epub 2017 Jun 20. PMID 28638000
- [Background] Ochentel O, Humphrey C, Pfeifer K. Efficacy of Exercise Therapy in Persons with Burnout. A Systematic Review and Meta-Analysis. J Sports Sci Med. 2018 Aug 14;17(3):475-484. eCollection 2018 Sep. PMID 30116121
- [Background] Tucker S, Farrington M, Lanningham-Foster LM, Clark MK, Dawson C, Quinn GJ, Laffoon T, Perkhounkova Y. Worksite Physical Activity Intervention for Ambulatory Clinic Nursing Staff. Workplace Health Saf. 2016 Jul;64(7):313-25. doi: 10.1177/2165079916633225. Epub 2016 May 3. PMID 27143144
- [Background] White MI, Dionne CE, Warje O, Koehoorn M, Wagner SL, Schultz IZ, Koehn C, Williams-Whitt K, Harder HG, Pasca R, Hsu V, McGuire L, Schulz W, Kube D, Wright MD. Physical Activity and Exercise Interventions in the Workplace Impacting Work Outcomes: A Stakeholder-Centered Best Evidence Synthesis of Systematic Reviews. Int J Occup Environ Med. 2016 Apr;7(2):61-74. doi: 10.15171/ijoem.2016.739. PMID 27112715
- [Background] Bridgland VME, Moeck EK, Green DM, Swain TL, Nayda DM, Matson LA, Hutchison NP, Takarangi MKT. Why the COVID-19 pandemic is a traumatic stressor. PLoS One. 2021 Jan 11;16(1):e0240146. doi: 10.1371/journal.pone.0240146. eCollection 2021. PMID 33428630
- [Background] Marcomini I, Agus C, Milani L, Sfogliarini R, Bona A, Castagna M. COVID-19 and post-traumatic stress disorder among nurses: a descriptive cross-sectional study in a COVID hospital. Med Lav. 2021 Jun 15;112(3):241-249. doi: 10.23749/mdl.v112i3.11129. PMID 34142675
- [Background] Tedeschi, R. G. & Calhoun, L. G. Posttraumatic growth: Conceptual foundations and empirical evidence. Psychological Inquiry 15, 1-18 (2004).
- [Background] National Center for Complementary and Integrative Health. (National Center for Complementary and Integrative Health, 2021).
- [Background] U.S. Department of Health and Human Services. Physical Activity Guidelines for Americans. 2nd edition edn, (Department of Health and Human Services, 2018).
- [Background] Linke SE, Gallo LC, Norman GJ. Attrition and adherence rates of sustained vs. intermittent exercise interventions. Ann Behav Med. 2011 Oct;42(2):197-209. doi: 10.1007/s12160-011-9279-8. PMID 21604068